CLINICAL TRIAL: NCT07179380
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled, Multicenter, Parallel Group Study to Evaluate the Efficacy and Safety of Treprostinil Palmitil Inhalation Powder in Participants With Pulmonary Hypertension Associated With Interstitial Lung Disease
Brief Title: Efficacy and Safety Study of Treprostinil Palmitil Inhalation Powder (TPIP) in Participants With Pulmonary Hypertension Associated With Interstitial Lung Disease (PH-ILD)
Acronym: PALM-ILD
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Insmed Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INS1009-311; 2025-521558-40-00 (Other: EU CT Number)
Record Dates: First submitted 2025-09-10; First posted 2025-09-17 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Pulmonary Hypertension; Interstitial Lung Disease
Keywords: pulmonary hypertension; interstitial lung disease
MeSH Terms: conditions — Hypertension, Pulmonary; Lung Diseases, Interstitial

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treprostinil Palmitil Inhalation Powder (Experimental): Participants will receive TPIP, once daily (QD), at a starting dose of 80 micrograms (μg) to maximum tolerated dose up to 1280 μg for 24 weeks.
  Interventions: Drug: Treprostinil Palmitil Inhalation Powder
- Placebo (Placebo Comparator): Participants will receive a placebo matching TPIP QD for 24 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Treprostinil Palmitil Inhalation Powder — Oral inhalation using a capsule-based dry powder inhaler device.
  Other Names: INS1009
  Arms: Treprostinil Palmitil Inhalation Powder
Drug: Placebo — Oral inhalation using a capsule-based dry powder inhaler device.
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the effect of 24-weeks of once daily treatment with TPIP versus placebo on exercise capacity in adults with PH-ILD.

ELIGIBILITY:
Inclusion Criteria

* Diagnosis of PH World Health Organisation (WHO) Group 3 associated with ILD [including but not limited to idiopathic interstitial pneumonia (IIP), chronic hypersensitivity pneumonitis (HSP), connective tissue disease-associated interstitial lung disease (CTD-ILD), combined pulmonary fibrosis and emphysema (CPFE)].
* Confirmation of fibrotic interstitial lung disease by centrally overread computed tomography (CT) scan performed at Screening or within prior 12 months.
* PH confirmed by right heart catheterization (RHC) at Screening or within 12 months prior to Screening, with the following hemodynamic findings:

  * Mean pulmonary arterial pressure (mPAP) >20 millimetre of mercury (mmHg) and
  * Pulmonary capillary wedge pressure (PCWP) of ≤15 mmHg and
  * Pulmonary vascular resistance (PVR) ≥4 wood units (WU).
* 6 Minute walking distance (6MWD) ≥100 and ≤500 meters at two 6MWTs at Screening performed at least 4 hours apart, with the difference between the 2 distances ≤15%.
* Participants receiving chronic medication for underlying disease (e.g., antifibrotic, immunomodulators, immunosuppressants, etc.) and/or phosphodiesterase 5 (PDE5) inhibitors, should be on this treatment for ≥90 days and on a stable dose for ≥30 days prior to Screening.
* Capable of giving signed informed consent as described in Section 10.1.5 which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion criteria

* Diagnosis of Pulmonary Hypertension WHO Groups 1, 2, 4, or 5, or subtypes of PH WHO Group 3 other than interstitial lung disease.
* Primary diagnosis of chronic obstructive pulmonary disease (COPD) and/or forced expiratory volume in 1 second (FEV1)/FVC <0.7 (based on screening or historical spirometry within the prior 6 months).
* Clinically significant left heart disease:

  * evidence of clinically significant left-sided valvular heart disease,
  * left ventricular failure with left ventricular ejection fraction (LVEF) <45%, or diagnosis of heart failure with preserved ejection fraction (HFpEF)
  * echocardiography findings at Screening suggestive for postcapillary PH
  * unstable ischemic heart disease
  * unstable arrhythmia, including uncontrolled atrial fibrillation (rate-controlled arrhythmia or paroxysmal atrial fibrillation is allowed)
* Evidence of chronic thromboembolic disease or recent (within 6 months of Screening) acute pulmonary embolism.
* Known hypersensitivity or contraindication to treprostinil or TPIP or TPIP formulation excipients (e.g., mannitol, leucine).
* Current use of cigarettes or e-cigarettes: An adult who has smoked at least 100 cigarettes in his or her lifetime and who currently smokes either every day or some days.
* Current use of inhaled marijuana, recreational or medical (current use defined as used at least one or more times during the past 30 days prior to Screening) or expected use during the study.
* Any other medical or psychological condition including relevant laboratory abnormalities at Screening that, in the opinion of the Investigator, suggest a new and/or insufficiently understood disease and/or may present an unreasonable risk to the study participant as a result of his/her participation in this clinical trial, may impede their ability complete the study or the study assessments or confound the outcomes of the trial.

Note: Other protocol defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Estimated)
Dates: Start 2026-01-07 (Actual); Primary Completion 2028-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in 6MWD Measured at Peak Exposure From Baseline to Week 24 | Baseline, Week 24

SECONDARY OUTCOMES:
Time From Randomization to First Clinical Worsening Over the 24-Week Treatment Period | Up to Week 24
Time From Randomization to First Major Morbidity or Mortality Event Over the 24-Week Treatment Period | Up to Week 24
Change From Baseline in N-Terminal Pro Hormone Brain Natriuretic Peptide (NT-proBNP) Plasma Concentration Over 24 Weeks | Baseline up to Week 24
Number of Participants With Greater Than or Equal to (>=) 30% Decrease in NT-proBNP or Who Maintained/Achieved Less Than (<) 300 Nanogram per Liter (ng/L) of NT-proBNP Level at Week 24 | At Week 24
Change in 6MWD Measured at Trough Exposure From Baseline to Week 22 | Baseline, Week 22
Change From Baseline in 6MWD Measured at Peak Exposure Over 20 Weeks | Baseline up to Week 20
Mean Change From Baseline in Living With Pulmonary Fibrosis (L-PF) Total Symptom Domain Score Over 24 Weeks | Baseline up to Week 24
Plasma Concentrations of Treprostinil Palmitil (TP) and Treprostinil (TRE) | Pre-dose and post-dose at multiple timepoints up to Week 24

CONTACTS AND LOCATIONS:
Locations (16):
- United States (4):
  - USA001, Santa Barbara, California
  - USA006, Naples, Florida
  - USA003, Bend, Oregon
  - USA008, Richmond, Virginia
- Georgia (3):
  - GEO004, Tbilisi
  - GEO003, Tbilisi
  - GEO001, Tbilisi
- Israel (3):
  - ISR003, Petah Tikva, Central District
  - ISR001, Haifa
  - ISR002, Jerusalem
- Japan (6):
  - JPN002, Narashino-shi, Chiba
  - JPN001, Sapporo, Hokkaido
  - JPN007, Yokohama, Kanagawa
  - JPN008, Kiyose, Tokyo
  - JPN003, Shibuya City, Tokyo
  - JPN005, Nagano

IPD SHARING:
Plan to Share IPD: No